CLINICAL TRIAL: NCT05806294
Title: Utilizing Canadian Digital Technology to Prevent and Manage Diabetes, Obesity, and Heart Disease in Patients Living With Congestive Obstructive Pulmonary Disease - A Single-arm Pilot Study
Brief Title: Digital Metabolic Rehabilitation COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Revive Wellness Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00116810
Record Dates: First submitted 2023-03-03; First posted 2023-04-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Syndrome; Chronic Obstructive Pulmonary Disease
Keywords: Web-based platform; Nutrition; Physical activity; Mindfulness; Primary care; Metabolic syndrome; COPD
MeSH Terms: conditions — Metabolic Syndrome; Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm pilot trial (Experimental): The Digital Metabolic Rehabilitation is a single-arm pilot trial that assesses Canadian Digital Technology's feasibility in preventing and managing MetS in patients living with COPD for a 6-month program.
  Interventions: Behavioral: Digital Metabolic Rehabilitation

INTERVENTIONS:
Behavioral: Digital Metabolic Rehabilitation — Digital Metabolic Rehabilitation combines two programs: The Canadian Health Advanced by Nutrition and Graded Exercise Protocol (CHANGE) and My Viva Plan (MVP). All participants receive free access to MVP and attend group video conferencing sessions with health professionals. After the 60-minute initial assessments with the dietitian and the kinesiologist, each participant has an individualized diet and exercise plan based on the intervention protocol built in MVP. Participants are split into groups of 20 based on physical ability and stage of COPD. Intervention has 3 phases. In phase 1, weekly videoconferences with the kinesiologist and dietitian and monthly sessions with psychologist and respiratory therapist are held for the first 3 months. Phase 2 lasts from months 4 to 6 and has biweekly videoconferences with health professionals. Phase 3 starts in month 6 and has monthly group sessions with health professionals.

SUMMARY:
People with Chronic Obstructive Pulmonary Disease (COPD) are at greater risk for Metabolic syndrome (MetS). Although the management of MetS will not cure COPD, it can beneficially impact health outcomes and quality of life through lifestyle modifications. The study aims to determine if using the Digital Metabolic Rehab program, which is based on preventive self-care and includes three key pillars of health: nutrition, fitness, and mindfulness, will be feasible to reduce or reverse MetS for individuals living with COPD.

DETAILED DESCRIPTION:
It is estimated that 50% of patients with Chronic Obstructive Pulmonary Disease (COPD) are at risk for having Metabolic Syndrome (MetS). While COPD is incurable, MetS can be reduced by diet and exercise. Yet, the evidence shows that lifestyle interventions with the self-management of health at home are low. Thus, the Canadian Health Advanced by Nutrition and Graded Exercise (CHANGE) protocol and My Viva Plan® (MVP) were created. CHANGE protocol is a personalized approach to nutrition and exercise modification supported by an interprofessional team in primary care settings. MVP is a digital Canadian self-care treatment program encompassing nutrition, fitness, and mindfulness. The investigators propose a 6-month Digital Metabolic Rehabilitation program using CHANGE protocol + MVP to guide diet and self-awareness in 50 individuals diagnosed with COPD and MetS. Assessments and measurements will be completed at baseline, 3 and 6 months. The study aims to determine the impact of the CHANGE protocol + MVP on reducing or reversing MetS for individuals living with COPD. This study will inform whether the Digital Metabolic Rehab program directly impacts health and wellness among patients with COPD and could become an essential tool for virtual, preventative self-care delivery in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18+)
* COPD stage 1 or 2
* Identified by their family doctor as having at least two out of five MetS factors
* Adjusted body mass index (BMI) between 26 to 40
* Able to provide written informed consent in English

Exclusion Criteria:

* Inability to speak, read or understand English
* Having a medical or physical condition that makes moderate-intensity physical difficult or unsafe
* Diagnosis of Type 1 diabetes mellitus or type 2 diabetes mellitus with proliferative diabetic retinopathy, nephropathy (serum creatine > 160 µmol/L), clinically significant neuropathy (defined as absent ankle jerks), severe hyperglycemia (fasting blood glucose > 11 mmol/L), or claudication symptoms
* Significant medical co-morbidities, including uncontrolled metabolic disorders (e.g., thyroid, renal, liver), COPD stages 3 or 4, heart failure stage D, stroke, and ongoing substance abuse, undergoing active treatment for cancer
* Clinically significant renal failure (.i.e., creatinine > 200 µmol/L)
* Diagnosis of psychiatric disorders that would limit the adequate ability to comply with the study protocol
* Unable or unwilling to use technology to meet with the healthcare team and My Viva Plan to manage self-care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Metabolic Syndrome | Change From baseline to month 3 and month 6
  Proportion of patients achieving reversal of Metabolic Syndrome (no longer meeting 3 of 5 diagnostic criteria)
Waist circumference | Change From baseline to month 3 and month 6
  Proportion of patients achieving reduction in waist circumference.
Blood pressure | Change From baseline to month 3 and month 6
  Proportion of patients achieving reduction in systolic and diastolic blood pressure. Systolic and diastolic blood pressure will be measured using a standard semi-automatic sphygmomanometer.

SECONDARY OUTCOMES:
Changes in body weight | From baseline to month 3 and month 6
  Changes in body weight will be measured using calibrated digital scale (Health o meter® Professional Remote Display, Sunbeam Products Inc., Fla., USA)
Changes in and body mass index (BMI) | From baseline to month 3 and month 6
  The intervention's ability to promote changes in BMI (weight and height will be combined to report BMI in kg/m^2)
Changes in fat mass | From baseline to month 3 and month 6
  Changes in fat mass (kg) by bioelectrical impedance analysis
Changes in phase angle | From baseline to month 3 and month 6
  Changes in phase angle is assessed by bioelectrical impedance analysis
Changes in fat-free mass | From baseline to month 3 and month 6
  Changes in fat-free mass (kg) by bioelectrical impedance analysis
Changes in muscle cross sectional area | From baseline to month 3 and month 6
  Changes in muscle cross sectional area (cm2) by ultrasound
Changes in muscle echogenicity | From baseline to month 3 and month 6
  Changes in muscle echogenicity by ultrasound
Changes in muscle strength | From baseline to month 3 and month 6
  Changes in muscle strength assessed by handgrip strength
Changes in physical performance | From baseline to month 3 and month 6
  Changes in physical performance assessed by 6-minute walk test
Changes in fitness assessment | From baseline to month 3 and month 6
  Changes in fitness test are assessed using the maximum number of partial curl-ups (up to 25) and push-ups performed in one minute.
Changes in flexibility test | From baseline to month 3 and month 6
  Changes in trunk flexion range of motion will be evaluated using inertial measuring units during bending in standing position.
Changes in resting energy expenditure | From baseline to month 3 and month 6
  Changes in resting energy expenditure assessed by indirect calorimetry

OTHER OUTCOMES:
Changes in quality of life parameters | From baseline to month 3 and month 6
  Changes in scores of quality of life are assessed by the Chronic Respiratory Questionnaire (CRQ). The Items are scaled in Numerical, 7-point modified Likert Scale. Higher scores indicate a better health-related quality of life
Changes in SF-12 score | From baseline to month 3 and month 6
  Changes in physical and mental well-being are assessed in 8 domains (physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health) by the Short Form 12 (SF-12).
Changes in cardiovascular disease risk | From baseline to month 3 and month 6
  Changes in cardiovascular disease risk by Prospective Cardiovascular Munster scores (PROCAM). PROCAM predicts cardiovascular risk in 10 years (<1% to > 40%). The higher the scores, the greater the cardiovascular risk
Well being changes | From baseline to month 3 and month 6
  Changes in well-being are assessed by the World Health Organization Well-Being Index (WHO-5). The raw scores are transformed to a score from 0 to 100, with lower scores indicating worse well-being
Mental health | From baseline to month 3 and month 6
  Mental health and depression are assessed by the Patient Health Questionnaire - 9 (PHQ-9). PHQ-9 score will be obtained by adding the score for each question (total points). Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively
Changes in psychosocial determinants of behavioral | From baseline to month 3 and month 6
  Physical Activity Readiness Questionnaire (PAR-Q+) will be used to assess the readiness of participants to engage in physical activity and determines any safety and possible risks that could be impacted by physical activity
Changes in hospital admissions rates for exacerbation of COPD | From baseline to month 6
  Exacerbation of COPD events is measured by outpatient visits, emergency room visits, and hospitalizations
Changes in hospital admissions rates for myocardial infarction events | From baseline to month 3 and month 6
  Myocardial infarction events are measured by outpatient visits, emergency room visits, and hospitalizations
Changes in hospital admissions rates for ischemic stroke events | From baseline to month 3 and month 6
  Ischemic stroke events are measured by outpatient visits, emergency room visits, and hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Doug Klein, MD, Principal Investigator — University of Alberta; Liam Collins, MS, Study Director — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CHANGE Alberta website — https://www.changealberta.net/
- See also: My Viva Plan website — https://discover.myvivaplan.com/